CLINICAL TRIAL: NCT02793583
Title: A Phase 2b Randomized Study to Assess the Efficacy and Safety of the Combination of Ublituximab + Umbralisib With or Without Bendamustine and Umbralisib Alone in Patients With Previously Treated Non-Hodgkin's Lymphoma
Brief Title: Study to Assess the Efficacy and Safety of Ublituximab + Umbralisib With or Without Bendamustine and Umbralisib Alone in Patients With Previously Treated Non-Hodgkins Lymphoma
Acronym: UNITY-NHL
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Strategic/Business Decision
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTX-TGR-205
Record Dates: First submitted 2016-05-23; First posted 2016-06-08 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Diffuse Large B-Cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma; Small Lymphocytic Lymphoma
Keywords: DLBCL; FL; MZL; MCL; SLL; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — ublituximab; umbralisib; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Umbralisib + Ublituximab (Experimental): Umbralisib oral daily dose in combination with Ublituximab intravenous administration
  Interventions: Biological: Ublituximab; Drug: Umbralisib
- Umbralisib (Experimental): Umbralisib oral daily dose
  Interventions: Drug: Umbralisib
- Umbralisib + Ublituximab + Bendamustine (Experimental): Umbralisib oral daily dose in combination with Ublituximab intravenous administration and Bendamustine intravenous administration
  Interventions: Biological: Ublituximab; Drug: Umbralisib; Biological: Bendamustine

INTERVENTIONS:
Biological: Ublituximab
  Other Names: TG-1101
  Arms: Umbralisib + Ublituximab; Umbralisib + Ublituximab + Bendamustine
Drug: Umbralisib
  Other Names: TGR-1202
Biological: Bendamustine
  Other Names: Treanda
  Arms: Umbralisib + Ublituximab + Bendamustine

SUMMARY:
Unity NHL - A Phase 2b Randomized Study to Assess the Efficacy and Safety of the Combination of Ublituximab + Umbralisib with or without Bendamustine and Umbralisib alone in Patients with Previously Treated Non-Hodgkin's Lymphoma

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of umbralisib monotherapy and the umbralisib + ublituximab (U2) combination in aggressive and indolent lymphomas and to also explore the U2 regimen in combination with bendamustine in the treatment of NHL (FL, SLL, MZL, DLBCL and MCL).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Non-Hodgkin's Lymphoma including Follicular, Mantle Cell Lymphoma and Marginal Zone Lymphoma
* Relapsed or refractory to prior standard therapy and subjects who are not candidates for high-dose therapy or autologous stem cell transplant
* MCL subjects with one or more lines of therapy including at least one BTK inhibitor (ibrutinib, acalabrutinib or zanibrutinib only)

Exclusion Criteria:

* Any major surgery, chemotherapy or immunotherapy within the last 21 days
* Evidence of hepatitis B virus, hepatitis C virus or known HIV infection
* Autologous hematologic stem cell transplant within 6 months of study entry. Prior Allogeneic hematologic stem cell transplant is excluded
* Prior therapy with a PI3K delta inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Every 8-12 weeks, up to 2 years

SECONDARY OUTCOMES:
Progression-Free Survival | From date of randomization until the date of first documented progression, assessed up through 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Owen A O'Connor, MD, PhD, Study Chair — Columbia University
Locations (147):
- United States (100):
  - TG Therapeutics Investigational Trial Site, Birmingham, Alabama
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Chandler, Arizona
  - TG Therapeutics Investigational Trial Site, Tucson, Arizona
  - TG Therapeutics Investigational Trial Site, Los Angeles, California
  - TG Therapeutics Investigational Trial Site, Orange, California
  - TG Therapeutics Investigational Trial Site, San Diego, California
  - TG Therapeutics Investigational Trial Site, Whittier, California
  - TG Therapeutics Investigational Trial Site, Aurora, Colorado
  - TG Therapeutics Investigational Trial Site, Denver, Colorado
  - TG Therapeutics Investigational Trial Site, Fort Collins, Colorado
  - TG Therapeutics Investigational Trial Site, Bridgeport, Connecticut
  - TG Therapeutics Investigational Trial Site, Newark, Delaware
  - TG Therapeutics Investigational Trial Site, Washington D.C., District of Columbia
  - TG Therapeutics Investigational Trial Site, Boca Raton, Florida
  - TG Therapeutics Investigational Trial Site, Fort Myers, Florida
  - TG Therapeutics Investigational Trial Site, Gainesville, Florida
  - TG Therapeutics Investigational Trial Site, Jacksonville, Florida
  - TG Therapeutics Investigational Trial Site, Miami, Florida
  - TG Therapeutics Investigational Trial Site, St. Petersburg, Florida
  - TG Therapeutics Investigational Trial Site, Tallahassee, Florida
  - TG Therapeutics Investigational Trial Site, Tampa, Florida
  - TG Therapeutics Investigational Trial Site, West Palm Beach, Florida
  - TG Therapeutics Investigational Trial Site, Albany, Georgia
  - TG Therapeutics Investigational Trial Site, Macon, Georgia
  - TG Therapeutics Investigational Trial Site, Marietta, Georgia
  - TG Therapeutics Investigational Trial Site, Chicago, Illinois
  - TG Therapeutics Investigational Trial Site, Decatur, Illinois
  - TG Therapeutics Investigational Trial Site, Evanston, Illinois
  - TG Therapeutics Investigational Trial Site, Harvey, Illinois
  - TG Therapeutics Investigational Trial Site, Maywood, Illinois
  - TG Therapeutics Investigational Trial Site, Niles, Illinois
  - TG Therapeutics Investigational Trial Site, Peoria, Illinois
  - TG Therapeutics Investigational Trial Site, Swansea, Illinois
  - TG Therapeutics Investigational Trial Site, Fort Wayne, Indiana
  - TG Therapeutics Investigational Trial Site, Indianapolis, Indiana
  - TG Therapeutics Investigational Trial Site, Westwood, Kansas
  - TG Therapeutics Investigational Trial Site, Louisville, Kentucky
  - TG Therapeutics Investigational Trial Site, Covington, Louisiana
  - TG Therapeutics Investigational Trial Site, Brewer, Maine
  - TG Therapeutics Investigational Trial Site, Baltimore, Maryland
  - TG Therapeutics Investigational Trial Site, Bethesda, Maryland
  - TG Therapeutics Investigational Trial Site, Columbia, Maryland
  - TG Therapeutics Investigational Trial Site, Towson, Maryland
  - TG Therapeutics Investigational Trial Site, Ann Arbor, Michigan
  - TG Therapeutics Investigational Trial Site, Duluth, Minnesota
  - TG Therapeutics Investigational Trial Site, Saint Louis Park, Minnesota
  - TG Therapeutics Investigational Trial Site, Columbia, Missouri
  - TG Therapeutics Investigational Trial Site, Kansas City, Missouri
  - TG Therapeutics Investigational Trial Site, St Louis, Missouri
  - TG Therapeutics Investigational Trial Site, Billings, Montana
  - TG Therapeutics Investigational Trial Site, Lincoln, Nebraska
  - TG Therapeutics Investigational Trial Site, Omaha, Nebraska
  - TG Therapeutics Investigational Trial Site, Lebanon, New Hampshire
  - TG Therapeutics Investigational Trial Site, Hackensack, New Jersey
  - TG Therapeutics Investigational Trial Site, Morristown, New Jersey
  - TG Therapeutics Investigational Trial Site, Mount Holly, New Jersey
  - TG Therapeutics Investigational Trial Site, Farmington, New Mexico
  - TG Therapeutics Investigational Trial Site, Buffalo, New York
  - TG Therapeutics Investigational Trial Site, New York, New York
  - TG Therapeutics Investigational Trial Site, Syracuse, New York
  - TG Therapeutics Investigational Trial Site, The Bronx, New York
  - TG Therapeutics Investigational Trial Site, Charlotte, North Carolina
  - TG Therapeutics Investigational Trial Site, Durham, North Carolina
  - TG Therapeutics Investigational Trial Site, Hickory, North Carolina
  - TG Therapeutics Investigational Trial Site, Kinston, North Carolina
  - TG Therapeutics Investigational Trial Site, Raleigh, North Carolina
  - TG Therapeutics Investigational Trial Site, Washington, North Carolina
  - TG Therapeutics Investigational Trial Site, Canton, Ohio
  - TG Therapeutics Investigational Trial Site, Cincinnati, Ohio
  - TG Therapeutics Investigational Trial Site, Cleveland, Ohio
  - TG Therapeutics Investigational Trial Site, Columbus, Ohio
  - TG Therapeutics Investigational Trial Site, Toledo, Ohio
  - TG Therapeutics Investigational Trial Site, Portland, Oregon
  - TG Therapeutics Investigational Trial Site, Springfield, Oregon
  - TG Therapeutics Investigational Trial Site, Camp Hill, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Philadelphia, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Providence, Rhode Island
  - TG Therapeutics Investigational Trial Site, Greenville, South Carolina
  - TG Therapeutics Investigational Trial Site, Sioux Falls, South Dakota
  - TG Therapeutics Investigational Trial Site, Watertown, South Dakota
  - TG Therapeutics Investigational Trial Site, Chattanooga, Tennessee
  - TG Therapeutics Investigational Trial Site, Kingsport, Tennessee
  - TG Therapeutics Investigational Trial Site, Knoxville, Tennessee
  - TG Therapeutics Investigational Trial Site, Memphis, Tennessee
  - TG Therapeutics Investigational Trial Site, Austin, Texas
  - TG Therapeutics Investigational Trial Site, Dallas, Texas
  - TG Therapeutics Investigational Trial Site, Fort Sam Houston, Texas
  - TG Therapeutics Investigational Trial Site, Houston, Texas
  - TG Therapeutics Investigational Trial Site, San Antonio, Texas
  - TG Therapeutics Investigational Trial Site, Tyler, Texas
  - TG Therapeutics Investigational Trial Site, Ogden, Utah
  - TG Therapeutics Investigational Trial Site, Blacksburg, Virginia
  - TG Therapeutics Investigational Trial Site, Newport News, Virginia
  - TG Therapeutics Investigational Trial Site, Olympia, Washington
  - TG Therapeutics Investigational Trial Site, Seattle, Washington
  - TG Therapeutics Investigational Trial Site, Spokane, Washington
  - TG Therapeutics Investigational Trial Site, Vancouver, Washington
  - TG Therapeutics Investigational Trial Site, Madison, Wisconsin
  - TG Therapeutics Investigational Trial Site, Wauwatosa, Wisconsin
- Australia (9):
  - TG Therapeutics Investigational Trial Site, Gosford, New South Wales
  - TG Therapeutics Investigational Trial Site, Wahroonga, New South Wales
  - TG Therapeutics Investigational Trial Site, Benowa, Queensland
  - TG Therapeutics Investigational Trial Site, South Brisbane, Queensland
  - TG Therapeutics Investigational Trial Site, Adelaide, South Australia
  - TG Therapeutics Investigational Trial Site, Heidelberg, Victoria
  - TG Therapeutics Investigational Trial Site, Nedlands, Western Australia
  - TG Therapeutics Investigational Trial Site, Netherlands, Western Australia
  - TG Therapeutics Investigational Trial Site, Gosford
- Israel (7):
  - TG Therapeutics Investigational Trial Site, Ashkelon
  - TG Therapeutics Investigational Trial Site, Beersheba
  - TG Therapeutics Investigational Trial Site, Haifa
  - TG Therapeutics Investigational Trial Site, Jerusalem
  - TG Therapeutics Investigational Trial Site, Nahariya
  - TG Therapeutics Investigational Trial Site, Petah Tikva
  - TG Therapeutics Investigational Trial Site, Tel Aviv
- Italy (5):
  - TG Therapeutics Investigational Trial Site, Bologna
  - TG Therapeutics Investigational Trial Site, Ferrara
  - TG Therapeutics Investigational Trial Site, Milan
  - TG Therapeutics Investigational Trial Site, Rome
  - TG Therapeutics Investigational Trial Site, Torino
- Poland (8):
  - TG Therapeutics Investigational Trial Site, Chorzów
  - TG Therapeutics Investigational Trial Site, Gdynia
  - TG Therapeutics Investigational Trial Site, Krakow
  - TG Therapeutics Investigational Trial Site, Lodz
  - TG Therapeutics Investigational Trial Site, Lublin
  - TG Therapeutics Investigational Trial Site, Słupsk
  - TG Therapeutics Investigational Trial Site, Warsaw
  - TG Therapeutics Investigational Trial Site, Wroclaw
- Slovakia (3):
  - TG Therapeutics Investigational Trial Site, Bratislava
  - TG Therapeutics Investigational Trial Site, Košice
  - TG Therapeutics Investigational Trial Site, Poprad
- South Korea (4):
  - TG Therapeutics Investigational Trial Site, Busan
  - TG Therapeutics Investigational Trial Site, Gyeonggi-do
  - TG Therapeutics Investigational Trial Site, Incheon
  - TG Therapeutics Investigational Trial Site, Seoul
- Spain (4):
  - TG Therapeutics Investigational Trial Site, Barcelona
  - TG Therapeutics Investigational Trial Site, Madrid
  - TG Therapeutics Investigational Trial Site, Salisbury
  - TG Therapeutics Investigational Trial Site, Valencia
- United Kingdom (7):
  - TG Therapeutics Investigational Trial Site, Cambridge
  - TG Therapeutics Investigational Trial Site, Denmark Hill
  - TG Therapeutics Investigational Trial Site, Leeds
  - TG Therapeutics Investigational Trial Site, Liverpool
  - TG Therapeutics Investigational Trial Site, London
  - TG Therapeutics Investigational Trial Site, Oxford
  - TG Therapeutics Investigational Trial Site, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared once the last patient visit has been completed

REFERENCES:
- [Derived] Fowler NH, Samaniego F, Jurczak W, Ghosh N, Derenzini E, Reeves JA, Knopinska-Posluszny W, Cheah CY, Phillips T, Lech-Maranda E, Cheson BD, Caimi PF, Grosicki S, Leslie LA, Chavez JC, Fonseca G, Babu S, Hodson DJ, Shao SH, Burke JM, Sharman JP, Law JY, Pagel JM, Miskin HP, Sportelli P, O'Connor OA, Weiss MS, Zinzani PL. Umbralisib, a Dual PI3Kdelta/CK1epsilon Inhibitor in Patients With Relapsed or Refractory Indolent Lymphoma. J Clin Oncol. 2021 May 20;39(15):1609-1618. doi: 10.1200/JCO.20.03433. Epub 2021 Mar 8. PMID 33683917